CLINICAL TRIAL: NCT05169554
Title: Beta-Lactam Containing Regimen for the Shortening of Buruli Ulcer Disease Therapy: Comparison of 8 Weeks Standard Therapy (Rifampicin Plus Clarithromycin) vs. 4 Weeks Standard Plus Amoxicillin/Clavulanate Therapy [RC8 vs. RCA4]
Brief Title: Beta-Lactam Containing Regimen for the Shortening of Buruli Ulcer Disease Therapy
Acronym: BLMs4BU
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fundacion Agencia Aragonesa para la Investigacion y Desarrollo (ARAID) (Other)
Collaborators: Universidad de Zaragoza (Other); Fondation Raoul Follereau (Unknown); Université d'Abomey-Calavi (Other); Instituto de Salud Carlos III (Other Government); Fundación Anesvad (Unknown); Tres Cantos Open Lab Foundation (Unknown); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TC281
Record Dates: First submitted 2021-11-22; First posted 2021-12-27 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Buruli Ulcer
Keywords: Buruli ulcer; Neglected tropical disease; Treatment shortening; Drug combination; Amoxicillin/clavulanate; Clinical trial; Pharmacokinetic analysis; Bacterial clearance study
MeSH Terms: conditions — Buruli Ulcer; Neglected Diseases | interventions — Clarithromycin; Therapeutics; Clavulanic Acid; WW Domain-Containing Oxidoreductase

STUDY DESIGN:
Intervention Model Description: BLMs4BU study is a Phase II, randomized, controlled open label non-inferiority, multi-centre trial, with two treatment arms:
  * Standard [RC8]: rifampicin plus clarithromycin (RC) therapy for 8 weeks; and
  * Investigational [RCA4]: standard (RC) plus amoxicillin/clavulanate (A) for 4 weeks.
  Randomization will be stratified by lesion category categories I, II or III, using a fixed block size within each strata.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RC8, Rifampicin plus Clarithromycin for 8 weeks (Active Comparator): Rifampicin plus Clarithromycin (RC) therapy for 8 weeks
  Interventions: Drug: Standard [RC8]: rifampicin plus clarithromycin (RC) therapy for 8 weeks.
- RCA4, Rifampicin plus Clarithromycin plus Amoxicillin/clavulanate for 4 weeks. (Experimental): Rifampicin plus Clarithromycin (RC) plus Amoxicillin/clavulanate (A) for 4 weeks.
  Interventions: Drug: Investigational [RCA4]: standard (RC) plus amoxicillin/clavulanate (A) for 4 weeks.

INTERVENTIONS:
Drug: Standard [RC8]: rifampicin plus clarithromycin (RC) therapy for 8 weeks. — Treatment will be rifampicin (600 mg, daily) and clarithromycin (500 mg, twice daily) for 8 weeks. On the posology, dosage for rifampicin and clarithromycin will be standardized according to patient body weight following WHO guidelines. In general, for a 60 kg adult dosage will be RIF, 10 mg/kg once daily and CLA, 7.5 mg/kg twice daily.
  Arms: RC8, Rifampicin plus Clarithromycin for 8 weeks
Drug: Investigational [RCA4]: standard (RC) plus amoxicillin/clavulanate (A) for 4 weeks. — On the posology, dosage for rifampicin and clarithromycin will be standardized according to patient body weight following WHO guidelines. In general, for a 60 kg adult dosage will be RIF, 10 mg/kg once daily and CLA, 7.5 mg/kg twice daily.
  Dosages for amoxicillin/clavulanate are calculated according to manufacturer indications:
  Dose of amoxicillin/clavulanate 1000/125 mg twice daily, which makes a total of 2000/250 mg/day, for patients over 40 kg, and 22.5/5.6 mg/kg twice daily, which makes a total of 45/11.25 mg/kg/day, for those equal and below 40 kg. For children, posology will be adapted to the age of the patient according to drug manufacturer indications. Frequency of AMX/CLV administration will match that of CLA, twice daily.
  Arms: RCA4, Rifampicin plus Clarithromycin plus Amoxicillin/clavulanate for 4 weeks.

SUMMARY:
Buruli ulcer (BU) is a skin Neglected Tropical Disease (NTD) that is caused by Mycobacterium ulcerans. It affects skin, soft tissues and bones causing long-term morbidity, stigma and disability. The greatest burden falls on children in sub-Saharan Africa. Treating BU requires 8-weeks with daily rifampicin and clarithromycin, wound care, and sometimes tissue grafting and surgery. Healing can take up to one year. Compliance is challenging due to socioeconomic determinants and may pose an unbearable financial burden to the household.

Recent studies led by members of this Consortium demonstrated that beta-lactams combined with rifampicin and clarithromycin are synergistic against M. ulcerans in vitro. Amoxicillin/clavulanate is oral, suitable for treatment in adults and children, and readily available with an established clinical pedigree. Its inclusion in a triple oral BU therapy has the potential of improving healing and shortening BU therapy.

The investigators propose a single blinded, randomized, controlled open label non-inferiority phase II, multi-centre trial in Benin with participants stratified according to BU category lesions and randomized in two oral regimens: (i) Standard [RC8]: rifampicin plus clarithromycin (RC) therapy for 8 weeks; and (ii) Investigational [RCA4]: standard (RC) plus amoxicillin/clavulanate (A) for 4 weeks. At least, a total of 140 patients will be recruited (70 per treatment arm), of which at least 132 will be PCR-confirmed. The primary efficacy outcome will be lesion healing without recurrence and without excision surgery 12 months after start of treatment (i.e. cure). A clinical expert panel assessing the need of excision surgery in both treatment arms will be blinded for treatment allocation in order to make objectives comparisons. Decision for excision surgery will be delayed to 14 weeks after initiation of antibiotic treatment. Secondary clinical efficacy outcomes include recurrence, treatment discontinuation and compliance rates, and the incidence of adverse effects, among others. In addition, two sub-studies will be performed: a pharmacokinetic (PK) analysis and a bacterial clearance study.

If successful, this study will create a new paradigm for BU treatment, which could inform changes in WHO policy and practice. This trial may also provide information on treatment shortening strategies for other mycobacterial infections, such as tuberculosis or leprosy.

ELIGIBILITY:
Inclusion Criteria:

All patients (both genders) with a new very likely or likely (WHO scoring criteria) clinical diagnosis of BU (all categories: I, II, III) and normal electrocardiogram (ECG) at baseline giving informed consent will be included in the study, as agreed by study site treatment team led by the lead clinicians.

Exclusion Criteria:

* Children < 5 years and adults >70 years.
* Children in foster care.
* Patients weighing less than 11 kilograms.
* Pregnancy positive (urine test: beta-HCG positive).
* Previous treatment of Buruli ulcer, tuberculosis or leprosy with at least one of the study drugs.
* Patients with diagnose leprosy or tuberculosis disease.
* Hypersensitivity to at least one of the study drugs or to any of the excipients.
* History of a severe immediate hypersensitivity reaction (e.g. anaphylaxis) to another beta-lactam agent (e.g. a cephalosporin, carbapenem or monobactam).
* History of jaundice/hepatic impairment due to amoxicillin/clavulanic acid or rifampicin.
* Patients with history of treatment with macrolide or quinolone antibiotics, anti-tuberculosis medication, or immuno-modulatory drugs including corticosteroids within one month.
* Patients currently receiving treatment with any drugs likely to interact with the study medications, i.e. anticoagulants, cyclosporine, phenytoin or phenobarbitone. Users of oral contraceptives should be notified that such contraceptive is less reliable if taken with rifampicin; additional (mechanical) contraceptive methods will be discussed with the study participant (Appendix 5).
* Patients with HIV co-infection.
* Patients with QTc prolongation >450 ms on ECG or on other medication known to prolong the QTc interval. In this case, if suspected of BU disease, patients will be offered 8-weeks rifampicin plus streptomycin therapy.
* Patients unable to take oral medication or having gastrointestinal disease likely to interfere with drug absorption.
* Patients with history or having current clinical signs of ascites, jaundice, myasthenia gravis, renal dysfunction (known or suspected), diabetes mellitus, and severe immune compromise, or evidence of tuberculosis, or leprosy; terminal illness (e.g., metastasized cancer), haematological malignancy, chronic liver disease, abnormal liver function test and coronary artery disease or any other condition that would preclude enrolment into the study in the study physician's opinion.
* Evidence of a clinically significant (as judged by the Investigator) condition or abnormality (other than the indication being studied) that might compromise safety or the interpretation of trial efficacy or safety endpoints
* Patients with known or suspected bowel strictures who cannot tolerate clarithromycin.
* Patients with a mental health condition that is likely to interfere with compliance with the study protocol in the opinion of the study physician.
* Patients (or parent/legal representative) who are not willing to give informed consent or withdrawal of consent.
* Specific exclusion criteria for the PK sub-study are patients less than 15 years old or less than 40 kg or with renal impairment with a creatinine level higher than the normal one in Benin (7-14 mg/L).

Ages: 5 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Cure rate, i.e. proportion of patients with complete lesion healing without recurrence and without excision surgery 12 months after treatment initiation, in the Per Protocol (PP) PCR+ population | 12 months after treatment initiation
  The PP PCR+ population includes those randomized patients with a clinical diagnosis of Very Likely BU or Likely BU, PCR+ and with no major violations of the protocol.

SECONDARY OUTCOMES:
Derive and compare the Area Under the Curve (AUC) (pharmacokinetic parameter) for RIF, CLA and AMX for the two groups (RC8 and RCA4) at steady-state. | Between week 1 and week 2 after treatment initiation
Derive and compare the trough concentration (Cτ) (pharmacokinetic parameter) for RIF, CLA and AMX for the two groups (RC8 and RCA4) at steady-state. | Between week 1 and week 2 after treatment initiation
Derive and compare the maximum observed drug concentration (Cmax) (pharmacokinetic parameter) for RIF, CLA and AMX for the two groups (RC8 and RCA4) at steady-state. | Between week 1 and week 2 after treatment initiation
Derive and compare the time to maximum observed drug concentration (tmax) (pharmacokinetic parameter) for RIF, CLA and AMX for the two groups (RC8 and RCA4) at steady-state. | Between week 1 and week 2 after treatment initiation
Derive and compare the elimination half-life (t1/2) (pharmacokinetic parameter) for RIF, CLA and AMX for the two groups (RC8 and RCA4) at steady-state. | Between week 1 and week 2 after treatment initiation
Characterize the POPPK in BU patients randomised on RCA4 and derive population PK arameters, such as apparent Clearance (CL/F), together with potential covariates of interest. | Between week 1 and week 2 after treatment initiation
  This will involve investigating inter- and intra-subject variability for RIF and AMX.
  The Pharmacokinetic Population (POPPK) is defined as the participants in the Safety Population (SP) who receive at least one dose of randomised study medication and have at least one evaluable PK sample. Participants will be analysed according to the treatment actually received.
Characterize the POPPK in BU patients randomised on RCA4 and derive population PK arameters, such as apparent Volume of distribution (V/F), together with potential covariates of interest. | Between week 1 and week 2 after treatment initiation
  This will involve investigating inter- and intra-subject variability for RIF and AMX.
  The Pharmacokinetic Population (POPPK) is defined as the participants in the Safety Population (SP) who receive at least one dose of randomised study medication and have at least one evaluable PK sample. Participants will be analysed according to the treatment actually received.
Characterize the POPPK in BU patients randomised on RCA4 and derive population PK arameters, such as Absorption Rate (Ka), together with potential covariates of interest. | Between week 1 and week 2 after treatment initiation
  This will involve investigating inter- and intra-subject variability for RIF and AMX.
  The Pharmacokinetic Population (POPPK) is defined as the participants in the Safety Population (SP) who receive at least one dose of randomised study medication and have at least one evaluable PK sample. Participants will be analysed according to the treatment actually received.
Rate of complete lesion healing without recurrence and without excision surgery, 12 months after start of treatment in the Intention-to-Treat Exposed (ITT-E) PCR+, PP Clinical Diagnose (CD), and ITT-E CD populations | 12 months after treatment initiation
  Intention To Treat Exposed (ITT-E) PCR + population:
  The ITT-E PCR+ population includes those randomized patients with a clinical diagnosis of Very Likely BU or Likely BU, PCR+ that have, at least, taken one dose of the study drugs. This population might include major violators of the protocol.
  Per Protocol (PP) Clinical Diagnose (CD) population:
  The PP CD population includes those randomized patients with a clinical diagnosis of Very Likely BU or Likely BU and with no major violations of the protocol. This population includes both PCR+ and PCR -.
  Intention To Treat Exposed (ITT-E) Clinical Diagnose (CD) population:
  The ITT-E CD population includes those randomized patients with a clinical diagnosis of Very Likely BU or Likely BU that have, at least, taken one dose of the study drugs. This population might include both PCR+ and PCR - and major violators of the protocol.
Rate of complete lesion healing without recurrence and without excision surgery 12 months after start of treatment by category (I, II & III) lesions analysis in all ITT-E and PP populations | 12 months after treatment initiation
  Intention-to-Treat Exposed (ITT-E): this population will consist of all randomized patients who receive at least one dose of randomized study medication. Patients will be assessed according to their randomized treatment, regardless of the treatment they receive.
  Per Protocol (PP): this population will consist of subjects in the ITT-E population who complete the study and are not major protocol violators.
Recurrence rate within 12 months of treatment initiation in all ITT-E and PP populations | Within 12 months of treatment initiation
  Intention-to-Treat Exposed (ITT-E): this population will consist of all randomized patients who receive at least one dose of randomized study medication. Patients will be assessed according to their randomized treatment, regardless of the treatment they receive.
  Per Protocol (PP): this population will consist of subjects in the ITT-E population who complete the study and are not major protocol violators.
Treatment discontinuation rate in all ITT-E and PP populations | Active comparator arm (RC8): 8 weeks; Experimental arm (RCA4): 4 weeks
  Intention-to-Treat Exposed (ITT-E): this population will consist of all randomized patients who receive at least one dose of randomized study medication. Patients will be assessed according to their randomized treatment, regardless of the treatment they receive.
  Per Protocol (PP): this population will consist of subjects in the ITT-E population who complete the study and are not major protocol violators.
Treatment compliance rate in all ITT-E and PP populations | Active comparator arm (RC8): 8 weeks; Experimental arm (RCA4): 4 weeks
  Intention-to-Treat Exposed (ITT-E): this population will consist of all randomized patients who receive at least one dose of randomized study medication. Patients will be assessed according to their randomized treatment, regardless of the treatment they receive.
  Per Protocol (PP): this population will consist of subjects in the ITT-E population who complete the study and are not major protocol violators.
Rate of paradoxical response within 12 months of treatment initiation in all ITT-E and PP populations | Within 12 months of treatment initiation
  Intention-to-Treat Exposed (ITT-E): this population will consist of all randomized patients who receive at least one dose of randomized study medication. Patients will be assessed according to their randomized treatment, regardless of the treatment they receive.
  Per Protocol (PP): this population will consist of subjects in the ITT-E population who complete the study and are not major protocol violators.
Median time to healing after treatment initiation in all ITT-E and PP populations | Within 12 months of treatment initiation until the date of healing time
  Intention-to-Treat Exposed (ITT-E): this population will consist of all randomized patients who receive at least one dose of randomized study medication. Patients will be assessed according to their randomized treatment, regardless of the treatment they receive.
  Per Protocol (PP): this population will consist of subjects in the ITT-E population who complete the study and are not major protocol violators.
Proportion of patients with reduction in lesion surface area within 12 months of treatment initiation in all ITT-E and PP populations | Within 12 months of treatment initiation
  Intention-to-Treat Exposed (ITT-E): this population will consist of all randomized patients who receive at least one dose of randomized study medication. Patients will be assessed according to their randomized treatment, regardless of the treatment they receive.
  Per Protocol (PP): this population will consist of subjects in the ITT-E population who complete the study and are not major protocol violators.
Interval between healing and recurrence within 12 months of treatment initiation in all ITT-E and PP populations | Within 12 months of treatment initiation
  Intention-to-Treat Exposed (ITT-E): this population will consist of all randomized patients who receive at least one dose of randomized study medication. Patients will be assessed according to their randomized treatment, regardless of the treatment they receive.
  Per Protocol (PP): this population will consist of subjects in the ITT-E population who complete the study and are not major protocol violators.
Incidence of all adverse events (AEs), Serious Adverse Events (SAE), Serious unexpected suspected adverse drug reactions (SUSAR) within 12 months of treatment initiation among treatment arms in all ITT-E and PP populations | Within 12 months of treatment initiation
  Intention-to-Treat Exposed (ITT-E): this population will consist of all randomized patients who receive at least one dose of randomized study medication. Patients will be assessed according to their randomized treatment, regardless of the treatment they receive.
  Per Protocol (PP): this population will consist of subjects in the ITT-E population who complete the study and are not major protocol violators.
Rate of median bacterial clearance among treatment arms in the bacterial clearance sub-study population | Within 8 weeks or 14 weeks after treatment initiation according to the healing time
Rate of patients with Buruli ulcer Functional Limitation Score (BUFLS) improvement within 12 months of treatment initiation among treatment arms in all ITT-E and PP populations | Within 12 months of treatment initiation
  Intention-to-Treat Exposed (ITT-E): this population will consist of all randomized patients who receive at least one dose of randomized study medication. Patients will be assessed according to their randomized treatment, regardless of the treatment they receive.
  Per Protocol (PP): this population will consist of subjects in the ITT-E population who complete the study and are not major protocol violators.

CONTACTS AND LOCATIONS:
Overall Officials: Santiago Ramón-García, Study Director — Fundacion Agencia Aragonesa para la Investigacion y Desarrollo (ARAID)
Locations (3):
- Benin (3):
  - Centre de Dépistage et de Traitement de l'Ulcère de Buruli (CDTUB) (Centers for Detection and Treatment of Buruli ulcer), Allada, Allada
  - Centre de Dépistage et de Traitement de l'Ulcère de Buruli (CDTUB) (Centers for Detection and Treatment of Buruli ulcer), Lalo, Lalo
  - Centre de Dépistage et de Traitement de l'Ulcère de Buruli (CDTUB) (Centers for Detection and Treatment of Buruli ulcer), Pobè, Pobè

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] O'Brien DP, Athan E, Blasdell K, De Barro P. Tackling the worsening epidemic of Buruli ulcer in Australia in an information void: time for an urgent scientific response. Med J Aust. 2018 Apr 16;208(7):287-289. doi: 10.5694/mja17.00879. No abstract available. PMID 29642808
- [Background] Revill WD, Morrow RH, Pike MC, Ateng J. A controlled trial of the treatment of Mycobacterium ulcerans infection with clofazimine. Lancet. 1973 Oct 20;2(7834):873-7. doi: 10.1016/s0140-6736(73)92005-9. No abstract available. PMID 4126917
- [Background] Espey DK, Djomand G, Diomande I, Dosso M, Saki MZ, Kanga JM, Spiegel RA, Marston BJ, Gorelkin L, Meyers WM, Portaels F, Deming MS, Horsburgh CR Jr. A pilot study of treatment of Buruli ulcer with rifampin and dapsone. Int J Infect Dis. 2002 Mar;6(1):60-5. doi: 10.1016/s1201-9712(02)90138-4. PMID 12044304
- [Background] Guarner J. Buruli Ulcer: Review of a Neglected Skin Mycobacterial Disease. J Clin Microbiol. 2018 Mar 26;56(4):e01507-17. doi: 10.1128/JCM.01507-17. Print 2018 Apr. PMID 29343539
- [Background] Thangaraj HS, Adjei O, Allen BW, Portaels F, Evans MR, Banerjee DK, Wansbrough-Jones MH. In vitro activity of ciprofloxacin, sparfloxacin, ofloxacin, amikacin and rifampicin against Ghanaian isolates of Mycobacterium ulcerans. J Antimicrob Chemother. 2000 Feb;45(2):231-3. doi: 10.1093/jac/45.2.231. PMID 10660507
- [Background] World Health Organization. Treatment of Mycobacterium ulcerans infection. 2012
- [Background] Boeree MJ, Diacon AH, Dawson R, Narunsky K, du Bois J, Venter A, Phillips PP, Gillespie SH, McHugh TD, Hoelscher M, Heinrich N, Rehal S, van Soolingen D, van Ingen J, Magis-Escurra C, Burger D, Plemper van Balen G, Aarnoutse RE; PanACEA Consortium. A dose-ranging trial to optimize the dose of rifampin in the treatment of tuberculosis. Am J Respir Crit Care Med. 2015 May 1;191(9):1058-65. doi: 10.1164/rccm.201407-1264OC. PMID 25654354
- [Background] Hu Y, Liu A, Ortega-Muro F, Alameda-Martin L, Mitchison D, Coates A. High-dose rifampicin kills persisters, shortens treatment duration, and reduces relapse rate in vitro and in vivo. Front Microbiol. 2015 Jun 23;6:641. doi: 10.3389/fmicb.2015.00641. eCollection 2015. PMID 26157437
- [Background] Omansen TF, Stienstra Y, van der Werf TS. Treatment for Buruli ulcer: the long and winding road to antimicrobials-first. Cochrane Database Syst Rev. 2018 Dec 17;12(12):ED000128. doi: 10.1002/14651858.ED000128. No abstract available. PMID 30556580
- [Background] Ramon-Garcia S, Gonzalez Del Rio R, Villarejo AS, Sweet GD, Cunningham F, Barros D, Ballell L, Mendoza-Losana A, Ferrer-Bazaga S, Thompson CJ. Repurposing clinically approved cephalosporins for tuberculosis therapy. Sci Rep. 2016 Sep 28;6:34293. doi: 10.1038/srep34293. PMID 27678056
- [Background] Arenaz-Callao MP, Gonzalez Del Rio R, Lucia Quintana A, Thompson CJ, Mendoza-Losana A, Ramon-Garcia S. Triple oral beta-lactam containing therapy for Buruli ulcer treatment shortening. PLoS Negl Trop Dis. 2019 Jan 28;13(1):e0007126. doi: 10.1371/journal.pntd.0007126. eCollection 2019 Jan. PMID 30689630
- [Background] Rolinson GN. Forty years of beta-lactam research. J Antimicrob Chemother. 1998 Jun;41(6):589-603. doi: 10.1093/jac/41.6.589. PMID 9687097
- [Background] Diacon AH, van der Merwe L, Barnard M, von Groote-Bidlingmaier F, Lange C, Garcia-Basteiro AL, Sevene E, Ballell L, Barros-Aguirre D. beta-Lactams against Tuberculosis--New Trick for an Old Dog? N Engl J Med. 2016 Jul 28;375(4):393-4. doi: 10.1056/NEJMc1513236. Epub 2016 Jul 13. No abstract available. PMID 27433841
- [Background] Ma Z, Lienhardt C, McIlleron H, Nunn AJ, Wang X. Global tuberculosis drug development pipeline: the need and the reality. Lancet. 2010 Jun 12;375(9731):2100-9. doi: 10.1016/S0140-6736(10)60359-9. Epub 2010 May 18. PMID 20488518
- [Background] Ramon-Garcia S, Ng C, Anderson H, Chao JD, Zheng X, Pfeifer T, Av-Gay Y, Roberge M, Thompson CJ. Synergistic drug combinations for tuberculosis therapy identified by a novel high-throughput screen. Antimicrob Agents Chemother. 2011 Aug;55(8):3861-9. doi: 10.1128/AAC.00474-11. Epub 2011 May 16. PMID 21576426
- [Background] Sarpong-Duah M, Frimpong M, Beissner M, Saar M, Laing K, Sarpong F, Loglo AD, Abass KM, Frempong M, Sarfo FS, Bretzel G, Wansbrough-Jones M, Phillips RO. Clearance of viable Mycobacterium ulcerans from Buruli ulcer lesions during antibiotic treatment as determined by combined 16S rRNA reverse transcriptase /IS 2404 qPCR assay. PLoS Negl Trop Dis. 2017 Jul 3;11(7):e0005695. doi: 10.1371/journal.pntd.0005695. eCollection 2017 Jul. PMID 28671942
- [Background] Kibadi K, Boelaert M, Fraga AG, Kayinua M, Longatto-Filho A, Minuku JB, Mputu-Yamba JB, Muyembe-Tamfum JJ, Pedrosa J, Roux JJ, Meyers WM, Portaels F. Response to treatment in a prospective cohort of patients with large ulcerated lesions suspected to be Buruli Ulcer (Mycobacterium ulcerans disease). PLoS Negl Trop Dis. 2010 Jul 6;4(7):e736. doi: 10.1371/journal.pntd.0000736. PMID 20625556
- [Background] Sarfo FS, Phillips RO, Zhang J, Abass MK, Abotsi J, Amoako YA, Adu-Sarkodie Y, Robinson C, Wansbrough-Jones MH. Kinetics of mycolactone in human subcutaneous tissue during antibiotic therapy for Mycobacterium ulcerans disease. BMC Infect Dis. 2014 Apr 15;14:202. doi: 10.1186/1471-2334-14-202. PMID 24731247
- [Background] Frimpong M, Agbavor B, Duah MS, Loglo A, Sarpong FN, Boakye-Appiah J, Abass KM, Dongyele M, Amofa G, Tuah W, Frempong M, Amoako YA, Wansbrough-Jones M, Phillips RO. Paradoxical reactions in Buruli ulcer after initiation of antibiotic therapy: Relationship to bacterial load. PLoS Negl Trop Dis. 2019 Aug 26;13(8):e0007689. doi: 10.1371/journal.pntd.0007689. eCollection 2019 Aug. PMID 31449522
- [Background] Roltgen K, Pluschke G. Buruli Ulcer: History and Disease Burden. 2019 Apr 30. In: Pluschke G, Roltgen K, editors. Buruli Ulcer: Mycobacterium Ulcerans Disease [Internet]. Cham (CH): Springer; 2019. Available from http://www.ncbi.nlm.nih.gov/books/NBK553836/ PMID 32091710
- [Background] Omansen TF, van der Werf TS, Phillips RO. Antimicrobial Treatment of Mycobacterium ulcerans Infection. 2019 Apr 30. In: Pluschke G, Roltgen K, editors. Buruli Ulcer: Mycobacterium Ulcerans Disease [Internet]. Cham (CH): Springer; 2019. Available from http://www.ncbi.nlm.nih.gov/books/NBK553822/ PMID 32091697
- [Background] Phillips RO, Robert J, Abass KM, Thompson W, Sarfo FS, Wilson T, Sarpong G, Gateau T, Chauty A, Omollo R, Ochieng Otieno M, Egondi TW, Ampadu EO, Agossadou D, Marion E, Ganlonon L, Wansbrough-Jones M, Grosset J, Macdonald JM, Treadwell T, Saunderson P, Paintsil A, Lehman L, Frimpong M, Sarpong NF, Saizonou R, Tiendrebeogo A, Ohene SA, Stienstra Y, Asiedu KB, van der Werf TS; study team. Rifampicin and clarithromycin (extended release) versus rifampicin and streptomycin for limited Buruli ulcer lesions: a randomised, open-label, non-inferiority phase 3 trial. Lancet. 2020 Apr 18;395(10232):1259-1267. doi: 10.1016/S0140-6736(20)30047-7. Epub 2020 Mar 12. PMID 32171422
- [Background] Wadagni AC, Barogui YT, Johnson RC, Sopoh GE, Affolabi D, van der Werf TS, de Zeeuw J, Kleinnijenhuis J, Stienstra Y. Delayed versus standard assessment for excision surgery in patients with Buruli ulcer in Benin: a randomised controlled trial. Lancet Infect Dis. 2018 Jun;18(6):650-656. doi: 10.1016/S1473-3099(18)30160-9. Epub 2018 Apr 5. PMID 29605498
- [Background] Sato T. A further look at the Cochran-Mantel-Haenszel risk difference. Control Clin Trials. 1995 Oct;16(5):359-61. doi: 10.1016/0197-2456(95)00004-6. No abstract available. PMID 8582154
- [Derived] Saez-Lopez E, Millan-Placer AC, Lucia A, Ramon-Garcia S. Amoxicillin/clavulanate in combination with rifampicin/clarithromycin is bactericidal against Mycobacterium ulcerans. PLoS Negl Trop Dis. 2024 Apr 4;18(4):e0011867. doi: 10.1371/journal.pntd.0011867. eCollection 2024 Apr. PMID 38573915
- [Derived] Johnson RC, Saez-Lopez E, Anagonou ES, Kpoton GG, Ayelo AG, Gnimavo RS, Mignanwande FZ, Houezo JG, Sopoh GE, Addo J, Orford L, Vlasakakis G, Biswas N, Calderon F, Della Pasqua O, Gine-March A, Herrador Z, Mendoza-Losana A, Diez G, Cruz I, Ramon-Garcia S. Comparison of 8 weeks standard treatment (rifampicin plus clarithromycin) vs. 4 weeks standard plus amoxicillin/clavulanate treatment [RC8 vs. RCA4] to shorten Buruli ulcer disease therapy (the BLMs4BU trial): study protocol for a randomized controlled multi-centre trial in Benin. Trials. 2022 Jul 8;23(1):559. doi: 10.1186/s13063-022-06473-9. PMID 35804454